CLINICAL TRIAL: NCT04791813
Title: Assessment of Maxillary Arch Depth and Width in a Group of Surgically Repaired Unilateral Cleft Lip and Palate Egyptian Children Versus Normal Children .A Cross Sectional Study
Brief Title: Assessment of Maxillary Arch Depth and Width in a Group of Surgically Repaired Unilateral Cleft Lip and Palate Children Versus Normal Children .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadir ahmed ali hassan, Principal investigator, Cairo University
Other Study IDs: H92
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: group of surgically treated unilateral cleft lip and palate Egyptian children aged 9_12years
  Interventions: Other: Alginate impressions , Photographic data and panoramic radiographs .
- Control group: group of healthy Egyptian children aged 9_12years
  Interventions: Other: Alginate impressions , Photographic data and panoramic radiographs .

INTERVENTIONS:
Other: Alginate impressions , Photographic data and panoramic radiographs . — Upper and lower alginate impressions will be poured and dental casts produced and converted to 3D digital cast using a 3D scanner-(3Shape )-the 3D data will be imported to a revers modeling software . Also Photographic data using Canon750 camera and panoramic radiographs to be taken.

SUMMARY:
The aim of the present study is to determine the effect of surgically repaired UCLP on dental arch dimensions and the need for orthodontic intervention in comparison with other healthy children , the presence of dental anomalies and the best possible standards of care among this group of Egyptian children.

DETAILED DESCRIPTION:
In arranging to distinguish and implement the best possible standards of care for UCLP children by the pediatric dental practitioner, evaluation of early treatment results after essential surgical repair of cleft lip and palate with respect to arch dimensions is fundamental. Although the dental arch dimensions for these children have been evaluated in previous studies , few examiners in Egypt handled this issue Due to racial contrasts in improvement of the dental arch and growth .The deficiency of data in Egypt tending to this insufficient assemble of children presents a gap that prevents the transport of fitting dental care to them. This is considered objective to fulfill this gap by spotting the most characteristics of dental arch dimensions in surgically repaired UCLP children and compares them with those of sound, coordinating, non-cleft.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative Egyptian children aging from ( 9-12) years.
* Medically free children.
* Children whose families accepts to participate in this study.
* Children with surgically repaired UCLP .

Exclusion Criteria:

* Children with previous untreated dental trauma.
* Children with previous orthodontic treatment
* Children with upper respiratory disease
* Children having any systemic diseases
* Intellectual disabilities or syndromes
* Congenital anomalies other than UCLP were excluded from the study .

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Egyptian children aging from 9-12 years old
Sampling Method: Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Inter canine maxillary arch width at the gingival level and 2. Inter molar maxillary arch Width at gingival level 3. Maxillary arch depth | Participants will be examined for once "day1"
  Inter canine maxillary arch width at the gingival level(between cusp tips of the right and left primary or permanent canines) 2. Inter molar maxillary arch Width at the gingival level(between mesio- buccul cusp tips of right and left first molars) 3. Maxillary arch depth( from the median point between central incisors to the tangent line between the distal surfaces of the second primary molars or mesial surfaces of first permanent molar.

SECONDARY OUTCOMES:
Percentage occurrence of dental abnormalities. | Participants will be examined for once " day 1"
  Percentage occurrence of hypodontia and other dental abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Hadir A Ali, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
Subject age, gender, maxillary arch dimensions, and dental anomalies found.